CLINICAL TRIAL: NCT04604834
Title: Autologous Platelet-rich Plasma (APRP) in the Treatment of Neurotrophic Keratopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Karim Mohamed-Noriega, Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OF14-004
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Neurotrophic Keratopathy
Keywords: Autologous PRP; Neurotrophic keratopathy; Autologous platelet-rich plasma

STUDY DESIGN:
Intervention Model Description: Subjects will be selected based on inclusion and exclusion criteria. A thorough ophthalmologic evaluation will be carried out before starting any treatment (baseline). Subjects will be randomly assigned to one of the treatment groups and receive the corresponding treatment for 4 weeks. At the end of week 4, subjects will switch treatment groups (crossover) and receive the new treatment for 4 more weeks. At the end of week 8, subjects will start the last treatment for 4 more weeks. Ophthalmologic evaluations will be performed every 4 weeks.
Masking Description: No blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PFAT first (Experimental): 1 eyedrop of PFAT every 2 hours in study eye.
  Interventions: Other: PFAT first
- APRP first (Experimental): 1 eyedrop of APRP every 2 hours in study eye.
  Interventions: Other: APRP first
- APRP+PFAT first (Experimental): 1 eyedrop of PFAT and APRP every 2 hours in study eye.
  Interventions: Other: PFAT first; Other: APRP first

INTERVENTIONS:
Other: PFAT first — Week 1 to week 4: one eyedrop of PFAT (preservative-free artificial tears) every 2 hours. Week 5 to week 8: one eyedrop of APRP (autologous plasma rich platelet) every 2 hours. Week 9 to week 12: one eyedrop of PFAT and APRP every 2 hours.
  Arms: APRP+PFAT first; PFAT first
Other: APRP first — Week 1 to week 4: one eyedrop of APRP every 2 hours. Week 5 to week 8: one eyedrop of PFAT every 2 hours. Week 9 to week 12: one eyedrop of PFAT and APRP every 2 hours.
  Arms: APRP first; APRP+PFAT first

SUMMARY:
Neurotrophic keratopathy (NK) is a condition where the cornea loses its capacity to feel pain and touch. This causes a decrease in the production of certain substances that maintain the integrity of the corneal epithelium (the most superficial layer that covers the cornea). As a result, the cornea cannot heal wounds as fast as it should and this could lead to corneal breakdown. This disease is chronic, meaning that it does not resolve quickly, and the treatments commonly used to manage it (such as artificial tears) take a long time to work, which makes it hard to follow doctor's orders. Autologous platelet-rich plasma is a substance that is obtained from the patient's own blood and it may contain those components that are missing in the tears of people with NK. The purpose of this experiment is to find out whether APRP+PFAT is better than APRP alone or PFAT alone in the treatment of NK. Participants will be randomly assigned to one of three groups: one group will start with APRP, other will start with PFAT and another with PFAT+APRP. The participants will receive each treatment for four weeks, and then the subjects will switch groups and use them for four weeks each (12 weeks total). Investigators will evaluate different parameters that will let us know if your condition is improving. These evaluations will be carried out every four weeks from the start to the end of the protocol. In case of intolerance or adverse effects, treatment will be discontinued.

DETAILED DESCRIPTION:
Neurotrophic keratopathy is characterized by impaired corneal sensitivity that results in a decrease in neurotrophic and epitheliotropic factors that are essential for proper corneal epithelial and ocular surface function. This neurotrophic state halts mitosis and epithelial turnover, which in turn slow down wound healing and lead to epithelial breakdown. Due to the chronicity of this disease, treatment adherence becomes a problem for patients; furthermore, results with conventional treatments such as preservative-free artificial tears are discouraging. Hematopoietic derivatives such as APRP may replace those missing neurotrophic factors and lead to epithelial healing in a faster and more comfortable manner. The objective of this study is to determine if APRP+PFAT is better than autologous platelet-rich plasma (APRP) or preservative-free artificial tears (PFAT) in the treatment of neurotrophic keratopathy. Subjects will be randomly assigned to one of three groups and treatment will be administered for four weeks. After this period, subjects will switch groups and receive the new treatment for four more weeks (cross-over). After this second period is completed, subjects will receive the last treatment for four more weeks. A thorough ophthalmologic evaluation will be performed before starting treatment and every four weeks until completion. Treatment will be discontinued if there are adverse effects or treatment intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

  * Neurotrophic keratopathy diagnosed by esthesiometry (defined as central corneal sensitivity ≤ 3cm using Cochet-Bonnet aesthesiometer).
  * Corneal erosions.
  * Neurotrophic keratopathy secondary to: diabetes mellitus, herpetic keratitis, microbial keratitis sequelae (bacteria, Acanthamoeba, fungi, herpes), limbal stem cell deficiency, chemical or thermic burn sequelae at least 3 months after the accident, ocular trauma with penetrating wound fixed at least 3 months before the trial, surgery carried out at least 3 month before the trial (including keratoplasty, laser in situ keratomileusis, phacoemulsification cataract surgery, extracapsular cataract extraction), adenoviral keratoconjunctivitis resolved at least 3 months the trial.

Exclusion Criteria:

* Patients diagnosed with:

  * Other ocular surface pathology presenting with corneal erosions but without corneal hyposensitivity.
  * Corneal epithelial defect with or without corneal hyposensitivity.
* Pregnant women, homeless, migrants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in corneal staining | from the beginning of the treatment and every 4 weeks until week 12.
  Change in corneal epithelial damage will be measured using corneal staining with fluorescein dye and the NEI grading scale.
Change in corneal sensitivity | from the beginning of the treatment and every 4 weeks until week 12.
  Change in corneal sensitivity will be measured using Cochet-Bonnet aesthesiometer.
Tear break-up time (TBUT) | from the beginning of the treatment and every 4 weeks until week 12.
  Tear break up time will be assessed using fluorescein dye, measuring break up time in seconds. A result >10 seconds will be considered normal, a result <10 seconds will be considered pathological.
Ocular Surface Disease Index (OSDI) | from the beginning of the treatment and every 4 weeks until week 12.
  Ocular surface symptoms will be assessed by the Ocular Surface Disease Index (OSDI). The OSDI questionnaire consists of 12 questions that assess dry eye symptoms and their effects on vision related function. The questionnaire is divided in 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients are asked to rate their responses on a 0 to 4 scale where 0 represents "none of the time", 1 "some of the time", 2 "half of the time", 3 "most of the time", and 4 "all of the time". The total score is calculated using the following formula: ([sum of scores for all questions answered x 100] / [total number of questions answered x 4]). Lower scores represent a better outcome.
Tear osmolarity. | from the beginning of the treatment and every 4 weeks until week 12.
  Tear osmolarity is one of tear inflammation biomarkers. Tear osmolarity will be performed with Tear Lab Osmolarity System, a result of 308 milliosmol (mOsm)/L or higher indicates pathological result.
Schirmer test with anesthesia | from the beginning of the treatment and every 4 weeks until week 12.
  Tear production will be measured by Schirmer test with anesthesia. The Schirmer test with anesthesia >15 mm is consider normal.
Quality of life questionnaire (National Eye Institute Visual Function Questionnaire-25) | from the beginning of the treatment and every 4 weeks until week 12.
  Quality of life as assessed by the National Eye Institute Visual Function Questionnaire (NEI VFQ-25). The NEI VFQ-25 questionnaire consists of 25 questions that assess the effect of visual impairment on the patient's quality of life. The 25-item questionnaire gives a score on a scale of 0 to 100, where 0 is the worst score and 100 is the best score. Higher scores represent a better outcome.
Best corrected visual acuity | from the beginning of the treatment and every 4 weeks until week 12.
  Best corrected visual acuity will be assessed using Snellen cards. Measurements will be converted to LogMar values for statistical analysis.
Frequency of adverse events. | from the beginning of the treatment and every 4 weeks until week 12.
  Frequency of adverse events will assessed for security and effectiveness of the treatment during the ophthalmic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Mohamed-Noriega, M.D., Principal Investigator — Departamento de Oftalmologia, Hospital Universitario Dr. Jose Eleuterio Gonzalez
Locations (1):
- Departamento de Oftalmologia, Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico